CLINICAL TRIAL: NCT05859893
Title: Therapeutic Melodies: How Classical Turkish Music Soothes Stress and Eases Loneliness - A Randomized Controlled Trial With Elders
Brief Title: Therapeutic Melodies: How Classical Turkish Music Soothes Stress and Eases Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Beycan Ekitli, PhD., Faculty member, lecturer, research associate, Ege University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: EgeTrial3
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Stress; Loneliness; COVID-19 Pandemic; Elderly
Keywords: livestream; music; tele-medicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The current 4-week randomized, single-blind factorial trial was conducted with a control group and one intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control (No Intervention)
- Intervention (Experimental): Behavioral: Interactive livestreamed classical Turkish music sessions with a professional music band.
  The sessions, which lasted approximately one and a half hours, twice a week, have been completed within one month.
  Interventions: Behavioral: Classical Turkish Music Sessions

INTERVENTIONS:
Behavioral: Classical Turkish Music Sessions — The participants attended an interactive livestreamed music performance. In selecting the mode, tempo, and songs to be performed, recommendations were obtained from the Applied Music Therapies Association, and the pieces with copyrighted recordings presented by the Edirne State Turkish Music Ensemble, under the leadership of the General Directorate of Fine Arts of the Ministry of Culture and Tourism. As part of the project, examples of traditional Turkish songs were presented to the elderly. The recommended genres and songs consist of vocal and instrumental works belonging to major and minor scales from the Classical Period, which spans from the 14th to the 20th century. In this respect an assembly of eight-musican consisting of five artists playing kanun, tanbur, ney, classical kemençe, and bendir, as well as two vocal soloists performed.
  Arms: Intervention

SUMMARY:
This study investigated the impact of traditional classical Turkish music as a telehealth intervention on reducing stress and loneliness among elderly individuals.

DETAILED DESCRIPTION:
The study was conducted at one of the Third Age University as a single-blind randomized and control-group experimental study. Elders were randomized into two main groups according to whether they lived alone or with someone. Interactive livestream musical interventions were performed for four weeks, in total eight sessions. The data of the study were collected three times with the Perceived Stress Scale and UCLA Loneliness Scale III in a pretest-posttest-follow-up test design (12th week after the posttest). Significance of difference tests, repeated variance analyses, and strength of influence tests were performed in dependent and independent groups with and without normal distribution.

The online-tool randomization method was utilized to apply simple randomization. Upon identifying the sample, it was initially segregated into two categories: individuals who resided alone and those who did not. The grouping of participants was carried out using an assignment method through a computer program, ensuring equivalence among research groups in terms of gender, stress, and loneliness. Following randomization, conformity of the groups' homogeneity and scales scores to normal distribution were examined with the Shapiro-Wilk test, skewness and kurtosis coefficients, histograms, and Levene's test of homogeneity of variance (p<0,05)

The study aimed to investigate the short and long-term effects of eight sessions of interactive livestreamed classic Turkish music performances on stress and loneliness during Covid-19 pandemic in elderly aged 65 and over who experiencing home isolation. The research hypotheses are as follows:

Perceived stress:

Hypothesis I, H1: Interactive livestream classical Turkish music sessions have a reducing effect on the mean scores of the Perceived Stress Scale.

i. There is a significant difference in the mean scores of the Perceived Stress Scale among intervention groups over time (pre-test, post-test, follow-up).

ii. There is a significant difference in the mean scores of the Perceived Stress Scale between intervention and control groups after the intervention in favor of the intervention group.

Loneliness:

Hypothesis II, H1: Interactive livestream classical Turkish music sessions have a reducing effect on the mean scores of the UCLA Loneliness Scale - III.

i. There is a significant difference in the mean scores of the UCLA Loneliness Scale - III among intervention groups over time (pre-test, post-test, follow-up).

ii. There is a significant difference in the mean scores of the UCLA Loneliness Scale - III between intervention and control groups after the intervention in favor of the intervention group.

For repeated measurements of score averages at different times within the same group, the homogeneity of variances was tested using the Levene Variance Homogeneity Assumption and Mauchly's Sphericity Assumption within the scope of Repeated Measures Analysis of Variance. When homogeneity could not be demonstrated, the Greenhouse-Geisser F value was used. For the control group with two-time measurements, the parametric repeated t-Test (Paired Samples t-Test) was used, assuming normal distribution.

To examine the significance of the difference in independent groups (intervention - control / intergroup) for repeated measurements at different times in assessing the effect size of the intervention, two-way repeated measures ANOVA (factorial ANOVA) was used. Since Mauchly's Sphericity Assumption was not met, the Greenhouse-Geisser F value was used, although the distribution was normal.

In the study, where the statistical significance level was accepted as p<0.05, effect size evaluations were made to test the statistical significance and confirm the practical applicability (in real conditions) of the findings. The effect size of the intervention was examined using partial eta squared (ηp2).

The data collection process was conducted thrice as pretest, posttest, and follow-up. The posttest was performed immediately after the completion of the 4-week intervention, whereas the follow-up measurements were obtained 12 weeks later. To apprise the volunteers about their respective groups and elucidate the application procedure, mobile appointments and virtual meetings were arranged.

ELIGIBILITY:
Inclusion Criteria:

* Registered for and attending their first years of lectures
* Aged higher than 65 year
* Able to use an interactive social media application via a computer, mobile phone or other electronic devices
* Participate willingly and voluntarily in the research.

Exclusion Criteria:

* Have a physical or sensory impairment that would affect the ability to listen to music (e.g., history of temporal brain damage, limb loss, hearing loss, etc.),
* Have a psychiatric diagnosis that would affect decision-making and orientation assessment abilities

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
The Perceived Stress Scale (first evaluation with posttest) | Through intervention completion, an average of 1 months
  Scale was developed by Cohen, Kamarck, and Mermelstein (1983), and adapted to Turkish culture by Eskin et al. (2013) to determine the potential effects of sample stress and loneliness perception on sociodemographic and musical tendencies. According to the psychometric adaptation study, criterion validity was ensured, with an internal consistency value of .84 and a test-retest reliability of .87. The scale, which consists of 14 items, is interpreted based on the total score and two sub-dimensions (Inadequate self-efficacy perception-ISPE and stress-discomfort perception-SDP). A high total score indicates a high perception of stress, inadequate coping strategies, and ineffective stress management. In this study, the Cronbach's alpha coefficient of the scale was 0.82.
The UCLA Loneliness Scale III (first evaluation with posttest) | Through intervention completion, an average of 1 months
  Scale is a widely used tool for assessing loneliness, which was developed by Russell et al. (1978). The psychometric properties of the UCLA Loneliness Scale III (UCLA-III) in Turkish culture were first investigated by Demir (1989). In this study, the 3rd revision of the scale developed by Durak and Senol Durak (2010) for Turkish culture was used. The scale consists of 20 items and is rated on a four-point Likert scale (1: Never - 4: Always). The total score ranges from 20 to 80, with higher scores indicating greater loneliness. In similar sample groups, the Cronbach's alpha coefficient of the scale was found to be 0.91, indicating high psychometric suitability (Kurt 2014). In the context of this study, the Chronbach's alpha coefficient of the scale is 0.93.
The Perceived Stress Scale (second evaluation with follow up) | Through intervention completion, an average of 3 months
  Scale was developed by Cohen, Kamarck, and Mermelstein (1983), and adapted to Turkish culture by Eskin et al. (2013) to determine the potential effects of sample stress and loneliness perception on sociodemographic and musical tendencies. According to the psychometric adaptation study, criterion validity was ensured, with an internal consistency value of .84 and a test-retest reliability of .87. The scale, which consists of 14 items, is interpreted based on the total score and two sub-dimensions (Inadequate self-efficacy perception-ISPE and stress-discomfort perception-SDP). A high total score indicates a high perception of stress, inadequate coping strategies, and ineffective stress management. In this study, the Cronbach's alpha coefficient of the scale was 0.82.
The UCLA Loneliness Scale III (second evaluation with follow up) | Through intervention completion, an average of 3 months
  Scale is a widely used tool for assessing loneliness, which was developed by Russell et al. (1978). The psychometric properties of the UCLA Loneliness Scale III (UCLA-III) in Turkish culture were first investigated by Demir (1989). In this study, the 3rd revision of the scale developed by Durak and Senol Durak (2010) for Turkish culture was used. The scale consists of 20 items and is rated on a four-point Likert scale (1: Never - 4: Always). The total score ranges from 20 to 80, with higher scores indicating greater loneliness. In similar sample groups, the Cronbach's alpha coefficient of the scale was found to be 0.91, indicating high psychometric suitability (Kurt 2014). In the context of this study, the Chronbach's alpha coefficient of the scale is 0.93.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Nursing, Izmır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Public data sharing is applicable to this article. It is planned to publish the research results in a high-impact journal in the field.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Approx 1 year after RCT registration.